CLINICAL TRIAL: NCT06043726
Title: Diagnostic Accuracy of Arterial-alveolar Oxygen Gradient in Low Risk Patients With Suspected Pulmonary Embolism
Acronym: DAGPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Franciscus Gasthuis (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-040
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Pulmonary Embolism
Keywords: A-a gradient
MeSH Terms: conditions — Pulmonary Embolism | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected PE: Patients with suspected pulmonary embolism
  Interventions: Diagnostic Test: Laboratory testing: D-dimeer and astrup

INTERVENTIONS:
Diagnostic Test: Laboratory testing: D-dimeer and astrup — Standard care: Laboratory result (D-dimer and astrup). CT scan for pulmonary embolism if indicated
  Other Names: CT-scan for pulmonary embolism

SUMMARY:
Introduction:

The diagnosis of pulmonary embolism (PE) is a challenge in the Emergency Department. D-dimer based diagnostic algorithms for PE have a very high sensitivity, but rely upon a vast amount of CT angiography and potentially unnecessary exposure to radiation. An accurate diagnostic algorithm that does not involve d-dimer testing might reduce this burden.

An abnormal Alveolar-arterial oxygen gradient (A-a gradient) seems to increase the chance of PE. However, a normal A-a gradient on its own does not exclude the diagnosis. In this paper, the accuracy of A-a gradient testing and a combination of Years criteria with A-a gradient testing will be assessed.

Methods:

This is a prospective, single center, observational study. All patients that present at our emergency department from September 2022 until September 2023 with a suspicion of pulmonary embolism will be analyzed for eligibility and included in the study after informed consent. The aim is to include at least 230 patients in the study.

Analysis: The primary outcome is the diagnostic accuracy of a YEARS and A-a gradient based algorithm for pulmonary embolism. The secondary outcome is the potential decrease in performed imaging in order to exclude pulmonary embolism.

Valorisation An accurate A-a gradient-based algorithm for pulmonary embolism in low risk patients will be a step towards an improved clinical risk score. We aim to reduce the amount of diagnostic imaging, i.e. CT-angiography. Meaning less, potentially unnecessary, exposure to radiation for the patient. Furthermore, it could lower healthcare costs by reducing expensive diagnostic imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patient with suspected pulmonary embolism
* Emergency department D-dimer result available
* Arterial blood gas available

Exclusion Criteria:

* Patients without documented oxygen suppletion durig blood gas measurement
* Patients without documented and insufficient data to calculate YEARS criteria
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients that present in our emergency department with suspicion of pulmonary embolism
Sampling Method: Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of a combination of a normal Alveolar-Arterial Oxygen Gradient with negative YEARS criteria in patients with suspected pumonary embolism | At submission in the Emergency Department

SECONDARY OUTCOMES:
How many CT-scans would have been avoided if the algorithm was used in normal practice | At submission in the Emergency Department

CONTACTS AND LOCATIONS:
Overall Officials: Sander Mol, Study Chair — Franciscus Gasthuis
Locations (1):
- Franciscus Gasthuis, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Hulle T, Cheung WY, Kooij S, Beenen LFM, van Bemmel T, van Es J, Faber LM, Hazelaar GM, Heringhaus C, Hofstee H, Hovens MMC, Kaasjager KAH, van Klink RCJ, Kruip MJHA, Loeffen RF, Mairuhu ATA, Middeldorp S, Nijkeuter M, van der Pol LM, Schol-Gelok S, Ten Wolde M, Klok FA, Huisman MV; YEARS study group. Simplified diagnostic management of suspected pulmonary embolism (the YEARS study): a prospective, multicentre, cohort study. Lancet. 2017 Jul 15;390(10091):289-297. doi: 10.1016/S0140-6736(17)30885-1. Epub 2017 May 23. PMID 28549662
- [Background] Kline JA, Courtney DM, Kabrhel C, Moore CL, Smithline HA, Plewa MC, Richman PB, O'Neil BJ, Nordenholz K. Prospective multicenter evaluation of the pulmonary embolism rule-out criteria. J Thromb Haemost. 2008 May;6(5):772-80. doi: 10.1111/j.1538-7836.2008.02944.x. Epub 2008 Mar 3. PMID 18318689
- [Background] McFarlane MJ, Imperiale TF. Use of the alveolar-arterial oxygen gradient in the diagnosis of pulmonary embolism. Am J Med. 1994 Jan;96(1):57-62. doi: 10.1016/0002-9343(94)90116-3. PMID 8304364
- [Background] Stein PD, Goldhaber SZ, Henry JW. Alveolar-arterial oxygen gradient in the assessment of acute pulmonary embolism. Chest. 1995 Jan;107(1):139-43. doi: 10.1378/chest.107.1.139. PMID 7632205
- [Background] Powrie RO, Larson L, Rosene-Montella K, Abarca M, Barbour L, Trujillo N. Alveolar-arterial oxygen gradient in acute pulmonary embolism in pregnancy. Am J Obstet Gynecol. 1998 Feb;178(2):394-6. doi: 10.1016/s0002-9378(98)80031-8. PMID 9500505
- [Background] Masotti L, Ceccarelli E, Cappelli R, Barabesi L, Forconi S. Arterial blood gas analysis and alveolar-arterial oxygen gradient in diagnosis and prognosis of elderly patients with suspected pulmonary embolism. J Gerontol A Biol Sci Med Sci. 2000 Dec;55(12):M761-4. doi: 10.1093/gerona/55.12.m761. PMID 11129400
- [Background] Overton DT, Bocka JJ. The alveolar-arterial oxygen gradient in patients with documented pulmonary embolism. Arch Intern Med. 1988 Jul;148(7):1617-9. PMID 3132902